CLINICAL TRIAL: NCT00783081
Title: Safety and Efficacy of K-134 for the Treatment of Intermittent Claudication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-134-2.01US
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Intermittent Claudication
Keywords: Intermittent Claudication; Peripheral Arterial Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — OPC 33509; Cilostazol; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- low dose K-134 (Experimental)
  Interventions: Drug: K-134
- mid dose K-134 (Experimental)
  Interventions: Drug: K-134
- high dose K-134 (Experimental)
  Interventions: Drug: K-134
- Comparator (Active Comparator)
  Interventions: Drug: Cilostazol 100 mg BID
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K-134 — K-134 is given as low dose mid dose and high dose tablets for 26 Weeks.
  Arms: high dose K-134; low dose K-134; mid dose K-134
Drug: Cilostazol 100 mg BID — Cilostazol 100mg BID for 26 weeks.
  Arms: Comparator
Drug: Placebo — Placebo BID for 26 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of K-134 for the treatment of intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

- Stable claudication symptoms

Exclusion Criteria:

* Lower extremity amputation
* Signs or symptoms of critical leg ischemia (CLI)
* Uncontrolled hypertension
* Tachycardia
* Poorly controlled diabetes
* Hypercholesterolemia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Improvement in peak walking time at 26 weeks | 26 Weeks

SECONDARY OUTCOMES:
Improvement in claudication onset time at 26 weeks | 26 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roger Morgan, M.D., FACS, Study Director — Kowa Research Institute, Inc.
Locations (42):
- United States (30):
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Los Angeles, California
  - Sacramento, California
  - Santa Rosa, California
  - Vista, California
  - Aurora, Colorado
  - Clearwater, Florida
  - Gulf Breeze, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Pensacola, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Aurora, Illinois
  - Chicago, Illinois
  - Hinsdale, Illinois
  - Indianapolis, Indiana
  - Auburn, Maine
  - St Louis, Missouri
  - Oklahoma City, Oklahoma
  - Danville, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Amarillo, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin
- Russia (12):
  - Gatchina
  - Irkutsk
  - Moscow
  - Novosibirsk
  - Pskov
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Sochi
  - Tomsk
  - Volgograd
  - Yaroslavl

REFERENCES:
- [Derived] Lewis RJ, Connor JT, Teerlink JR, Murphy JR, Cooper LT, Hiatt WR, Brass EP. Application of adaptive design and decision making to a phase II trial of a phosphodiesterase inhibitor for the treatment of intermittent claudication. Trials. 2011 May 25;12:134. doi: 10.1186/1745-6215-12-134. PMID 21612611